CLINICAL TRIAL: NCT02645851
Title: RApid Fluid Volume EXpansion (RVE) in Critically Ill Patients With Acute Circulatory Failure After the Initial Phase of Resuscitation. A Single-center, Open-label, Randomized Study Comparing 3 Strategies of RVE in Orléans, France.
Brief Title: RApid Fluid Volume EXpansion in Patients in Shock After the Initial Phase of Resuscitation.
Acronym: RAVEXO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties for the recruitment of patients
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRO-2015-02; 2015-A00311-48 (Registry Identifier: IDRCB (Identifiant de Recherche et Collections Biologiques))
Record Dates: First submitted 2015-12-27; First posted 2016-01-05 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Shock; Hypovolemia
Keywords: Fluid Therapy; Plasma Substitutes; Fluid Balance
MeSH Terms: conditions — Shock; Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- "PLR-induced SV changes" based strategy (Experimental): During the intervention period (i.e., within 120 hrs following inclusion), every time a fluid bolus is deemed necessary to improve the patient's cardiac output, the final decision to administer or not the fluid bolus will be determined by the percentage changes in Stroke Volume (SV) observed during a 1-min Passive Leg Raising test: Administration of the fluid bolus if SV changes ≥10%, or no administration otherwise. Measurement of beat-to-beat stroke volume by intraarterial pulse contour analysis using the PiCCO system (Pulsion, Germany) will be used to assess stroke volume changes. Per protocol inclusion criteria, patients will be carrying central venous and artery catheters.
  Interventions: Drug: fluid bolus; Device: PiCCO system (Pulsion, Germany); Device: Vascular pressure transducers (Edwards Life Science, USA); Other: Passive Leg Raising test
- "PLR-induced PP changes" based strategy (Experimental): During the intervention period (i.e., within 120 hrs following inclusion), every time a fluid bolus is deemed necessary to improve the patient's cardiac output, the final decision to administer or not the fluid bolus will be determined by the percentage changes in Pulse Pressure (PP) observed during a 1-min Passive Leg Raising test: Administration of the fluid bolus if PP changes ≥10%, or no administration otherwise. We will perform measurement of intraarterial blood pressure using vascular pressure transducers (Edwards Life Science, USA). Per protocol inclusion criteria, patients will be carrying central venous and artery catheters.
  Interventions: Drug: fluid bolus; Device: Vascular pressure transducers (Edwards Life Science, USA); Other: Passive Leg Raising test
- Usual Care (Other): During the intervention period (i.e., within 120 hrs following inclusion), every time a fluid bolus is deemed necessary to improve the patient's cardiac output, the fluid bolus will be administered without measurement of any predictive index of fluid responsiveness. Per protocol inclusion criteria, patients will be carrying central venous and artery catheters.
  Interventions: Drug: fluid bolus; Device: Vascular pressure transducers (Edwards Life Science, USA)

INTERVENTIONS:
Drug: fluid bolus — Administration of the fluid bolus if deemed clinically necessary, OR if deemed clinically necessary AND PLR-induced SV or PP changes ≥10%, depending of the Arm the patient is assigned to
  Other Names: vascular volume expansion
Device: PiCCO system (Pulsion, Germany) — During the intervention period (from inclusion to the 120th hour), every time a fluid bolus is deemed necessary, fluid responsiveness will be assessed by Stroke Volume changes obtained at 1 min of a Passive Leg Raising (PLR) test (fluid will be given if PLR-induced stroke volume change is over 10%; in case stroke volume change is below 10%, fluid will not be given and need for fluid reassessed after a short period of time, as in usual care)
  Arms: "PLR-induced SV changes" based strategy
Device: Vascular pressure transducers (Edwards Life Science, USA) — During the intervention period (from inclusion to the 120th hour), every time a fluid bolus is deemed necessary, fluid responsiveness will be assessed by Pulse Pressure changes obtained at 1 min of a Passive Leg Raising (PLR) test (fluid will be given if PLR-induced Pulse Pressure change is over 10%; in case Pulse Pressure change is below 10%, fluid will not be given and need for fluid reassessed after a short period of time, as in usual care)
Other: Passive Leg Raising test — Passive elevation of the legs of the patient, and lying down of the trunk (if patient is in the semi-recumbent position), preferably using electric bed. If not available, elevation of the legs by an assistant to a 45 degrees angle. Effects of Passive Leg Raising on Pulse Pressure or on Stroke Volume are used to assess fluid responsiveness in patients suffering from shock states.
  Other Names: Passive elevation of the legs of the patient.
  Arms: "PLR-induced PP changes" based strategy; "PLR-induced SV changes" based strategy

SUMMARY:
Rapid volume expansion using repeated intravenous fluid boluses is a very common intervention performed in the intensive care unit (ICU) in the early days of resuscitation of patients with shock. Once passed the initial phase of resuscitation, the fluid boluses administered fail to effectively increase the patients' cardiac output in about 50% of cases. Pulse pressure changes or stroke volume changes induced by a Passive Leg Raising (PLR) test have acceptable/good ability to predict fluid responsiveness (in terms of cardiac output change) and may be systematically used in patients with persistent shock with the aim of limiting the total amount of fluid administered to patients by avoiding undue fluid boluses. One may suppose that such a volume expansion management policy could impact morbidity and mortality of shocked patients. Among the predictive indices available in clinical practice, the PLR test has the advantages of being usable regardless of the patients' respiratory status and cardiac rhythm. Changes in left ventricular stroke volume during the PLR test perform better that changes in pulse pressure to predict fluid responsiveness. However, in counterpart, pulse pressure changes during PLR can be assessed without the need of other hemodynamic exploration such central venous pressure measurement or cardiac output monitoring. The investigators hypothesized that strategies using either stroke volume changes or pulse pressure changes induced by the PLR test to decide wether a fluid bolus clinically deemed indicated should or should not be administered, may limit the amount of fluid received by the patients during the first 5 days of shock, improve their oxygenation index, and shorten the time passed under mechanical ventilation, as compared to a "liberal" strategy (usual care) that does not use predictive indices of fluid responsiveness.

DETAILED DESCRIPTION:
A pilot, single-center, randomized, open-label, 3 parallel groups clinical trial with 1:1:1 assignment of interventions, comparing outcomes between patients with persistent shock assigned to either 1) the "Volume expansion guided by PLR-induced changes in Stroke Volume" strategy, or 2) the "Volume expansion guided by PLR-induced changes in Pulse Pressure" strategy, or 3) to usual care (i.e., without the use of any predictive index of fluid responsiveness). Patients in shock (either of septic, cardiac or other origin) will be included once passed the first hours of resuscitation. The time window for inclusion will be from 6 to 24 hours after the beginning of resuscitation, a delay necessary to ensure that initial hypovolemia has been fully compensated.

The randomization will be stratified according to the presumed origin of shock (cardiac, septic, or other) and according to the PaO2/FiO2 ratio (<200 or ≥ 200 mmHg).

The randomly assigned intervention will be used during the first 5 days of shock (120 hours).

ELIGIBILITY:
Pre-eligibility criteria:

* Patients presenting on Intensive Care Unit (ICU) admission or later during their ICU stay with arterial hypotension (Mean arterial pressure [MAP]<65mmHg or systolic arterial pressure [SAP]< 90 mmHg at least two times over a 15-minute interval), regardless of the method used to measure blood pressure (invasive or non invasive),
* Or patients already receiving continuous iv vasopressor therapy on ICU admission, regardless of the blood pressure level, will be considered as potential candidates for inclusion in the study, depending on his/her clinical evolution after 6 to 24 hours of care according to current guidelines for shock management.
* In case arterial hypotension is present and/or the patient is already receiving continuous iv vasopressor at ICU admission, the date and time of admission will be considered as the time of shock onset (H0).
* In case arterial hypotension occurs after ICU admission, the date and time of the first episode of hypotension will be considered as the time of shock onset (H0).

Inclusion Criteria:

* Patients will be eligible for inclusion if 6 hours after H0 (and before H24) all the following conditions are present:
* Informed consent obtained (or emergency inclusion possible when legal representatives and patient's family are not present, as allowed by the Ethic Committee and by the French Law)
* Persistence of arterial hypotension (as defined above) or continuous iv infusion of norepinephrine
* Patient under invasive mechanical ventilation
* At least one of the following conditions is present
* Alteration of consciousness
* Mottling skin
* Cyanosis of the extremities despite SaO2>90%
* Oliguria defined as urine output below 0.5ml/kg of actual body weight over at least 1 hour
* Arterial lactate > 2 mmol/L
* ScvO2 < 70%
* Central venous (internal jugular or subclavian) or femoral venous catheter in place
* Arterial catheter in place

Exclusion Criteria:

1. Shock began more than 24 hours ago
2. Age < 18 yrs.
3. Pregnancy
4. Uncontrolled haemorrhage
5. Intra-aortic balloon counterpulsation in place
6. Patient under veno-arterial extracorporeal membrane oxygenation (V-A ECMO)
7. Cardiogenic pulmonary oedema during the past 24 hours
8. Patient equipped with a cardiac output monitoring device
9. Brain death
10. Moribund patient
11. Traction of a lower limb
12. Amputated lower limb above the ankle level
13. Documented intra-abdominal hypertension

13. Cardiac arrest motivating ICU admission or cardiac arrest since admission 14. Patient without social security number 15. Consent refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio changes | from inclusion to the 24th hour after inclusion

SECONDARY OUTCOMES:
ventilator free days | ventilator free days between inclusion and the 28th day
  Every complication related to intravenous or arterial catheters inserted during the intensive care unit stay will be recorded
Catheter-related complications | from inclusion to the date of intensive care unit discharge, an average of 10 days
  Every complication related to intravenous or arterial catheters inserted during the intensive care unit stay will be recorded
Fluid balance | from inclusion to the 7th day
Immediate respiratory tolerance of fluid bolus (Yes or No) | at each fluid bolus administered during the intervention period (from inclusion to 120 hours later)
  Definition of immediate respiratory tolerance: SpO2 drops by less than 3% AND respiratory rate increase by less than 20% between before and after fluid bolus AND no occurrence of clinical pulmonary edema.
mortality rate | at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Boulain, MD, Principal Investigator — Centre Hospitalier Régional d'Orléans, France
Locations (1):
- Centre Hospitalier Régional d'Orléans, France, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annane D, Sebille V, Charpentier C, Bollaert PE, Francois B, Korach JM, Capellier G, Cohen Y, Azoulay E, Troche G, Chaumet-Riffaud P, Bellissant E. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA. 2002 Aug 21;288(7):862-71. doi: 10.1001/jama.288.7.862. PMID 12186604
- [Background] Annane D, Sebille V, Duboc D, Le Heuzey JY, Sadoul N, Bouvier E, Bellissant E. Incidence and prognosis of sustained arrhythmias in critically ill patients. Am J Respir Crit Care Med. 2008 Jul 1;178(1):20-5. doi: 10.1164/rccm.200701-031OC. Epub 2008 Apr 3. PMID 18388358
- [Background] Antonelli M, Levy M, Andrews PJ, Chastre J, Hudson LD, Manthous C, Meduri GU, Moreno RP, Putensen C, Stewart T, Torres A. Hemodynamic monitoring in shock and implications for management. International Consensus Conference, Paris, France, 27-28 April 2006. Intensive Care Med. 2007 Apr;33(4):575-90. doi: 10.1007/s00134-007-0531-4. PMID 17285286
- [Background] Benes J, Chytra I, Altmann P, Hluchy M, Kasal E, Svitak R, Pradl R, Stepan M. Intraoperative fluid optimization using stroke volume variation in high risk surgical patients: results of prospective randomized study. Crit Care. 2010;14(3):R118. doi: 10.1186/cc9070. Epub 2010 Jun 16. PMID 20553586
- [Background] Boulain T, Achard JM, Teboul JL, Richard C, Perrotin D, Ginies G. Changes in BP induced by passive leg raising predict response to fluid loading in critically ill patients. Chest. 2002 Apr;121(4):1245-52. doi: 10.1378/chest.121.4.1245. PMID 11948060
- [Background] Boulain T, Garot D, Vignon P, Lascarrou JB, Desachy A, Botoc V, Follin A, Frat JP, Bellec F, Quenot JP, Mathonnet A, Dequin PF; Clinical Research in Intensive Care and Sepsis Group. Prevalence of low central venous oxygen saturation in the first hours of intensive care unit admission and associated mortality in septic shock patients: a prospective multicentre study. Crit Care. 2014 Nov 6;18(6):609. doi: 10.1186/s13054-014-0609-7. PMID 25529124
- [Background] Boulain T, Boisrame-Helms J, Ehrmann S, Lascarrou JB, Bougle A, Chiche A, Lakhal K, Gaudry S, Perbet S, Desachy A, Cabasson S, Geneau I, Courouble P, Clavieras N, Massanet PL, Bellec F, Falquet Y, Reminiac F, Vignon P, Dequin PF, Meziani F. Volume expansion in the first 4 days of shock: a prospective multicentre study in 19 French intensive care units. Intensive Care Med. 2015 Feb;41(2):248-56. doi: 10.1007/s00134-014-3576-1. Epub 2014 Dec 2. PMID 25447804